CLINICAL TRIAL: NCT07094607
Title: The Effect of Ecological Intelligence and Ecological Anxiety on Organic Food Consumers' Sustainable Nutrition Behaviors
Brief Title: The Impact of Ecological Intelligence and Anxiety on Sustainable Nutrition
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: Sedef Güngör-Atılım-02
Record Dates: First submitted 2025-05-20; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Ecological Anxiety; Ecological Intelligence; Sustainable Dietary Preferences
Keywords: eco-anxiety; ecological intellegence; organic food consumers; sustainable nutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group (participants consuming organic food): It will consist of individuals between the ages of 18-65 who live in Ankara and declare that they have been consuming organic food for at least six months.
- Control group (participants who do not consume organic food): Individuals who live in Ankara, who do not declare that they consume organic food or who have consumed organic food for less than 6 months and who have similar characteristics with the study group between the ages of 18-65 will be included.

SUMMARY:
Environmental problems such as climate change, loss of biodiversity and depletion of natural resources threaten sustainable living and human health. In order to cope with these threats, individuals' environmental sensitivity should be increased and sustainable lifestyles should be encouraged. In this context, ecological intelligence refers to the ability of individuals to transform environmental knowledge into sustainable behaviors, while ecological anxiety defines the anxiety against environmental threats and may lead individuals to environmentally friendly consumption behaviors. In particular, organic food consumption is considered as a reflection of both ecological intelligence and ecological anxiety. Individuals who prefer organic products make more conscious choices with the aim of reducing environmental impacts and eating healthy. Accordingly, ecological intelligence and ecological anxiety stand out as important factors affecting individuals' sustainable and healthy eating behaviors.

Aim: This study aims to examine the effects of ecological intelligence and ecological concern on sustainable eating behaviors in organic food consumers.

Expected Results of the Study:

This project aims to examine the effects of ecological intelligence and ecological anxiety levels on the sustainable eating behaviors of organic food consumers. The results may show that increased levels of environmental knowledge and concern may reflect positively on sustainable dietary choices and that these individuals are more conscious in their organic food choices. It may also contribute to the development of strategies to promote ecological awareness and environmentally friendly consumption behaviors.

DETAILED DESCRIPTION:
Introduction:

Environmental problems such as climate change, declining biodiversity and depletion of natural resources pose a major threat to sustainable living and human health. In order to cope with these environmental problems, increasing the environmental awareness of individuals is vital for the adoption of sustainable lifestyles. Concern about environmental problems can contribute to individuals' orientation towards conscious consumption behaviors. In this context, the concept of ecological intelligence refers to individuals' ability to acquire environmental knowledge and transform this knowledge into sustainable behaviors. Ecological intelligence improves individuals' ability to both minimize their environmental impact and make healthy life choices. It is thought that the level of ecological intelligence can contribute to individuals' sustainable and healthy eating behaviors and help them to reduce their environmental impact.

Ecological anxiety is a concept that describes the anxiety individuals feel about climate change and other environmental threats. Ecological anxiety can lead individuals to adopt environmentally friendly consumption decisions, which in turn promotes sustainable food choices such as organic food consumption. Organic food consumers generally tend to make more conscious choices in terms of environmental sustainability and health. These individuals seek to protect both their health and the environment by turning to environmentally friendly production methods and products free from chemical additives.

In this context, organic food consumption is seen in the dietary habits of individuals with high environmental awareness as a reflection of ecological intelligence. Organic agriculture has the potential to limit environmental degradation by reducing the use of chemical fertilizers and pesticides and contributes to sustainable food consumption. It is reported that organic food consumers prefer foods that are free from chemical additives and produced with natural methods in order to ensure environmental sustainability and develop healthy eating habits. In addition, research has also shown that individuals with high levels of ecological anxiety increase their organic food consumption due to their environmental concerns. This reinforces individuals' willingness to make sustainable food choices and the impact of ecological intelligence.

This study aims to examine the relationship between ecological intelligence levels of organic food consumers and their sustainable and healthy eating behaviors. Understanding how the ecological intelligence levels of organic food consumers affect their sustainable eating habits is of great importance in terms of promoting environmentally friendly lifestyles. The findings of the study may contribute to the development of strategies for individuals to develop healthier and sustainable eating habits by improving their environmental awareness. In addition, by filling the gap in the literature on the relationship between organic food consumers' ecological intelligence levels and dietary behaviors, it will contribute to the creation of a solid knowledge base for increasing awareness of sustainable food consumption.

Method:

Research Design This research will be conducted with a cross-sectional case-control study design and will examine the differences between individuals who consume organic food (study group) and individuals who do not consume organic food (control group). This design allows for a comparative examination of the relationships between ecological intelligence, ecological anxiety and sustainable eating behaviors between the two groups.

Research Sample The research sample will consist of 64 participants who consume organic food (study group) and 64 participants who do not consume organic food (control group), totaling at least 128 people. It is planned to include people with similar age, gender and socioeconomic characteristics from both groups. For the "study group", the sample will consist of individuals aged 18-65 living in Ankara and declaring that they have been consuming organic food for at least six months. For the "control group", the sample will consist of individuals aged 18-65 who live in Ankara, do not declare that they consume organic food and have similar characteristics with the study group.

Data Collection Process Participants will be informed about the purpose of the study and it will be stated that confidentiality principles will be followed, consent will be obtained from the voluntary participants and the scales will be applied to both groups in the same order. For this, individuals will fill out "Informed voluntary consent forms". Individuals who will participate in the study will be reached through social media, online organic food groups or organic markets. Data will be collected from the participants through face-to-face survey applications.

Data Collection Tools Demographic information of the participants (age, gender, height, weight, presence of chronic diseases, etc.) and information about their eating habits will be obtained with a questionnaire form.

Ecological Intelligence Scale: It was developed to measure individuals' environmental knowledge, awareness and ability to transform it into sustainable behaviors. The original version of the scale was created by Daniel Goleman based on the theoretical framework for the concept of ecological intelligence. The Turkish adaptation of the scale and its validity and reliability study was carried out by Okur-Berberoğlu, and it was confirmed as a suitable tool for measuring environmental awareness and sustainable living behaviors of individuals in Turkey. This scale will be used in the project to determine the environmental sensitivity levels of individuals and to examine the relationship between sustainable eating behaviors and ecological intelligence.

Eco-Anxiety Scale: The Eco-Anxiety Scale is based on the concept of "eco-anxiety" developed by Hogg et al. to measure the level of anxiety and worry felt by individuals in the face of environmental problems. The original version of the scale focuses on assessing the psychological effects of global ecological threats such as climate change and environmental crises. The validity and reliability study of this scale in Turkey was conducted by Uzun et al. In this project, the Eco-anxiety Scale will be used to determine the ecological anxiety levels of organic food consumers and to evaluate the effects of this anxiety on sustainable eating behaviors and ecological intelligence. In this context, it will help to analyze the reflection of individuals' concerns about environmental problems on conscious consumption and sustainable living habits.

Sustainable and Healthy Eating Behaviors Scale: It is a scale developed to assess individuals' behaviors towards sustainability and healthy eating habits. This scale was first prepared by Żakowska-Biemans et al. to determine sustainable eating habits. It was adapted into Turkish and its validity and reliability study was conducted by Köksal et al. Within the scope of the project, the Sustainable and Healthy Eating Behaviors Scale will be used to assess the sustainable eating behaviors of organic food consumers. This scale will be associated with variables such as ecological intelligence and ecological anxiety by analyzing the environmental sensitivity of individuals through their dietary preferences.

Expected Results of the Study:

This project aims to examine the effects of ecological intelligence and ecological anxiety levels on the sustainable eating behaviors of organic food consumers. The results may show that increased levels of environmental knowledge and concern may reflect positively on sustainable dietary preferences and that these individuals are more conscious in their organic food choices. It may also contribute to the development of strategies to promote ecological awareness and environmentally friendly consumption behaviors.

ELIGIBILITY:
Inclusion Criteria:

* To reside in Ankara
* Being between the ages of 18-65

Exclusion Criteria:

* Being outside the 18 - 65 age range
* Not residing in Ankara

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals between 18 - 65 years of age, residing in Ankara
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in sustainable nutrition behaviours according to ecological intelligence level | Up to three month
  'Ecological Intelligence Scale for Adults' will be used to measure the ecological intelligence of individuals. There are 12 statements in this scale. The statements in the scales are asked on a 5-point Likert scale. The minimum score that can be obtained from this scale is 12 and the maximum score is 60. The higher the score, the higher the level of ecological anxiety. There is no cut-off value. 'Sustainable and Healthy Eating Behaviours Scale' will be used to measure sustainable eating behaviours. The scale consists of a total of 32 questions and is scored on a 7-point Likert scale. The scale has a total of 7 subgroups. These are evaluated by factor scoring. Then, the total score of the scale is obtained by calculating the average of the scores obtained for 7 subgroups. The minimum value obtained from the total score is 1 and the maximum value is 7. Both subgroup and total score correlation will be analysed to determine the change between the two.
The change in sustainable nutrition behaviours of individuals according to their ecological anxiety levels | Up to three month
  'Eco-anxiety Scale' will be used to measure the ecological anxiety of individuals. There are 13 statements in this scale. The statements in the scales are asked on a 4-point Likert scale. The minimum score that can be obtained from this scale is 0 and the maximum score is 39. The higher the score, the higher the level of ecological anxiety. There is no cut-off value. 'Sustainable and Healthy Eating Behaviours Scale' will be used to measure sustainable eating behaviours. The scale consists of 32 questions in total and is scored on a 7-point Likert scale. The scale has a total of 7 subgroups. These are evaluated by factor scoring. Then, the total score of the scale is obtained by calculating the average of the scores obtained for 7 subgroups. The minimum value obtained from the total score is 1 and the maximum value is 7. Both subgroup and total score correlation will be analysed to determine the change between the two.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)